CLINICAL TRIAL: NCT00712764
Title: Role of Adenosine in the Control of Choroidal Blood Flow During Changes in Ocular Perfusion Pressure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Michael Wolzt, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-011206
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Ocular Physiology; Microcirculation
Keywords: Adenosine; Choroidal blood flow; Suction cup
MeSH Terms: interventions — Adenosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Adenosine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adenosine
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Autoregulation is the ability of a vascular bed to maintain blood flow despite changes in perfusion pressure. For a long time it had been assumed that the choroid is a strictly passive vascular bed, which shows no autoregulation. However, recently several groups have identified some autoregulatory capacity of the human choroid. In the brain and the retina the mechanism behind autoregulation is most likely linked to changes in transmural pressure. In this model arterioles change their vascular tone depending on the pressure inside the vessel and outside the vessel. In the choroid, several observations argue against a direct involvement of arterioles. However, the mechanism behind choroidal autoregulation remains unclear. Adenosine, an endogenous purine metabolic end product with a potent vasodilatory effect on multiple vascular beds, leads to an increase in retinal and choroidal vessel diameter. The present study aims to investigate whether adenosine plays a role in choroidal autoregulation during a decrease in ocular perfusion pressure, which will be achieved by an increase in intraocular pressure.

Pressure/flow relationships will be investigated in the absence and presence of adenosine.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
choroidal pressure-flow relationship | 2 hours at 2 study days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Schmidl D, Weigert G, Dorner GT, Resch H, Kolodjaschna J, Wolzt M, Garhofer G, Schmetterer L. Role of adenosine in the control of choroidal blood flow during changes in ocular perfusion pressure. Invest Ophthalmol Vis Sci. 2011 Jul 29;52(8):6035-9. doi: 10.1167/iovs.11-7491. PMID 21697134